CLINICAL TRIAL: NCT04385095
Title: A Randomised Double-blind Placebo-controlled Trial to Determine the Safety and Efficacy of Inhaled SNG001 (IFN-β1a for Nebulisation) for the Treatment of Patients With Confirmed SARS-CoV-2 Infection
Brief Title: Trial of Inhaled Anti-viral (SNG001) for SARS-CoV-2 (COVID-19) Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Synairgen Research Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SG016
Record Dates: First submitted 2020-04-24; First posted 2020-05-12 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: SARS-CoV-2
Keywords: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Randomised double-blind placebo-controlled
  Pilot phase - 100 patients randomised in the hospital setting, 120 patients randomised in the home setting.
  Pivotal phase - estimated at an additional 100 to 300 patients per arm, but the actual number will be determined after the data review at the end of the Pilot phase
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SNG001 (Active Comparator): inhalation using the I-neb device.
  Interventions: Drug: SNG001
- Placebo (Placebo Comparator): inhalation using the I-neb device.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SNG001 — SNG001 via inhalation
  Arms: SNG001
Drug: Placebo — Placebo via inhalation
  Arms: Placebo

SUMMARY:
SNG001 is an inhaled drug that contains a antiviral protein called interferon beta (IFN-β). IFN-β in produced in the lungs during viral lung infections. It has been shown that older people and people with some chronic diseases have an IFN-β deficiency. Many viruses inhibit IFN-β as part of their strategy to evade the immune system.

Addition of IFN-β in vitro protects lung cells from viral infection. IFN-β protects cells against the MERS and SARS coronaviruses (close relatives of SARS-CoV-2, the virus that causes COVID-19).

SNG001 is an inhaled formulation of interferon beta-1a it is currently in Phase II clinical trials for COPD patients.

Synairgen has conducted randomised placebo controlled clinical trials of SNG001 involving >200 asthma and COPD patients. These trials have shown that SNG001 has:

* been well tolerated during virus infections
* enhanced antiviral activity in the lungs (measured in sputum and blood samples)
* provided significant lung function benefit over placebo in asthma in two Phase II trials.

Synairgen believes SNG001 could help prevent worsening or accelerate recovery of severe lower respiratory tract illness in COVID-19 patients.

Patients who are in hospital or non-hospitalised but are a high risk groups (e.g. elderly or diabetics) will be invited to take part in the trial. The patient would receive either SNG001 or placebo once daily for 14 days. The severity of the patients condition would be recorded on a scale developed by the World Health Organisation and the patient would be asked questions about their breathlessness, cough and sputum every day, as well as assess their general medical condition and safety.

The study will start as a Pilot phase where 100 patients will be randomised in the hospital setting and a 120 patients randomised in the home setting.

Once each of the Pilot phases are complete, a Pivotal phase will be conducted. It is estimated that the size of each of the Pivotal phases (hospital and home) will be around 100 to 300 patients per arm. The actual number will be determined after the data review at the end of each of the Pilot phases.

If SNG001 proves to be beneficial it would be a major breakthrough for the treatment of COVID-19.

ELIGIBILITY:
Inclusion Criteria:

1. A. Hospital setting: positive virus test for SARS-CoV-2 using RT-PCR, or positive point-of-care viral infection test in the presence of strong clinical suspicion of SARS-CoV-2 infection.

   B. Home setting: positive virus test for SARS-CoV-2 using a molecular assay e.g. RT-PCR in the presence of strong clinical suspicion of SARS-CoV-2 infection.
2. Male or female, ≥18 years of age (hospital setting) or ≥50 years of age (home setting) at the time of consent.
3. A. Hospital setting: patients admitted to hospital due to the severity of their COVID 19 disease OR

   B. Home setting: non-hospitalised patients from high-risk groups, defined as ≥65-years of age, or ≥50 years of age and with any of the following risk factors:
   * Arterial hypertension
   * Cardiovascular disease
   * Diabetes mellitus
   * Chronic lung disease
   * Chronic kidney disease (eGFR <60 mL/min/1.73m2)
   * Chronic liver disease
   * Immunodeficiency due to a serious illness or medication
   * Cerebrovascular disease
   * Malignancy (except basal cell carcinoma) diagnosed in the last 5 years
   * Body Mass Index ≥30 who present with clinical symptoms consistent with COVID-19:
   * High temperature and/or
   * New, continuous cough.
   * Loss or change to sense of smell and/or taste
4. Provide informed consent.
5. A. Hospital setting: hospitalised female patients must be ≥1 year post-menopausal, surgically sterile, or using an acceptable method of contraception.

B. Home setting: non-hospitalised female patients must be ≥1 year post-menopausal or surgically sterile.

Exclusion Criteria:

1. > 24 hours after confirmation of SARS-CoV-2 infection by a molecular assay e.g. RT-PCR test (hospital and home settings) or >24 hours after a positive point-of-care viral infection test (hospital setting only). This criterion does not apply to patients in the hospital setting who had their positive RT-PCR test for SARS-CoV-2 performed prior to hospitalisation.
2. ≥ 8 days from onset of COVID-19 symptoms (cough and/or fever and/or loss or change to sense of smell and/or taste; home setting only).
3. Any condition, including findings in the patients' medical history or in the pre-randomisation study assessments that in the opinion of the Investigator, constitute a risk or a contraindication for the participation of the patient into the study or that could interfere with the study objectives, conduct or evaluation.
4. Current or previous participation in another clinical trial where the patient has received a dose of an Investigational Medicinal Product (IMP) containing small molecules within 30 days or 5 half-lives (whichever is longer) prior to entry into this study or containing biologicals within 3 months prior to entry into this study.
5. Ventilated or in intensive care.
6. Inability to use a nebuliser with a mouthpiece.
7. History of hypersensitivity to natural or recombinant IFN-β or to any of the excipients in the drug preparation.
8. Females who are breast-feeding, lactating, pregnant or intending to become pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2020-03-16 (Actual); Primary Completion 2021-02-17 (Actual); Study Completion 2021-11-16 (Actual)

PRIMARY OUTCOMES:
Ordinal Scale for Clinical Improvement | Day 1 to Days 15 and 28
  Change in condition measured using the Ordinal Scale for Clinical Improvement during the dosing period - minimum of 0 (patient is well) to a maximum of 8 (death)

SECONDARY OUTCOMES:
Progression to pneumonia (hospital setting only) | Day 2 to Day 28
  Progression to pneumonia as diagnosed by chest x-ray, if no pneumonia is present at time of enrolment
Progression to pneumonia (hospital setting only) | Day 1 to Day 28
  Evolution of pneumonia, as diagnosed by chest x-ray, if pneumonia is present at time of enrolment
Time to clinical improvement (hospital setting only) | Time to hospital discharge OR Time to NEWS2 of ≤ 2 maintained for 24 hours
  Time to clinical improvement
National Early Warning Score 2 (NEWS2) assessment of acute-illness severity (hospital setting only) | Day 1 to Day 28
  NEWS2 assessment of acute-illness severity on a scale of 0 ( being well) up to 24 (requiring emergency response)
Changes in daily breathlessness, cough and sputum scale (BCSS) | Day 1 to Day 28 (and Day 60 and 90 home setting only)
  Changes in daily breathlessness, cough and sputum scale (BCSS) on a scale of 0 (no symptoms) up to 4 (severe symptoms)
Safety and tolerability - blood pressure (hospital setting only) | Day 1 to Day 15
  Looking at blood pressure measured in mmHg
Safety and tolerability - heart rate | Day 1 to Day 15
  Looking at heart rate measured in beats per minute
Safety and tolerability - temperature | Day 1 to Day 15
  Looking at temperature measured in degrees Celsius
Safety and tolerability - respiratory rate (hospital setting only) | Day 1 to Day 15
  Looking at respiratory rate measure in breaths per minute
Safety and tolerability - oxygen saturation | Day 1 to Day 15
  Looking at oxygen levels measured in a %
Safety and tolerability - adverse events | Day 1 to Day 28
  Looking at adverse events (numbers and terms)
Safety and tolerability - concomitant medications | Day 1 to Day 28
  Looking at concomitant medications given during treatment
Time to clinical improvement (home setting only) | Day 1 to Day 15
  Temperature ≤37.8 °C AND COVID-19 symptoms (breathing, cough, sputum, muscle aches, headache, fatigue, sore throat, loss or change to sense of smell and taste, rhinorrhoea and anorexia) all rated as absent or mild
Time to improvement of COVID-19 symptoms (home setting only). | Day 1 to Day 28 and Day 60 and 90
  Time to improvement of COVID-19 symptoms (fever, breathing, cough, sputum, muscle aches, headache, fatigue, sore throat, loss or change to sense of smell and/or taste, rhinorrhoea and anorexia)
Time to self-reported recovery (home setting only) | Day 2 to Day 15 and Day 28, 60 and 90
  Time to self-reported recover
Self-reported daily rating of overall feeling of wellness (home setting only). | Day 1 to Day 28 and Day 60 and 90
  Self-reported daily rating of overall feeling of wellness scale from 1 (the worst you can imagine) to 10 (the best you can imagine)
Quality of life measured using EQ-5D-5L (home setting only). | Day 1 to Day 28 and Day 60 and 90
  Quality of life measured using EQ-5D-5L - 5 questions where minimum score is 1 (best outcome) to 5 (worst outcome), visual analogue scale is also included for this 100 is best health you can imagine to 0 worst health you can imagine
Virus clearance/load (if samples are available) | Day 1 to Day 28
  Time to virus clearance and viral load
Blood and sputum biomarkers (if samples are available). | Day 1 to Day 28
  Blood and sputum biomarkers
Contact with health services (home setting only) | Day 1 to Day 28
  Contact with health services
Consumption of antibiotics (home setting only) | Day 1 to Day 28
  Consumption of antibiotics
General Anxiety Disorder 7 (home setting only) | Day 60 and 90
  Assessment of anxiety - score of 0 (best) to 3 (worst)
Patient Health Questionnaire - 9 | Day 60 and 90
  Assessment of mental health - score of 0 (best) to 3 (worst)
FACIT Fatigue Scale | Day 60 and 90
  Assessment of Fatigue - score of 0 (best) to 4 (worst)
Nottingham Extended Activities of Daily Living Scale | Day 60 and 90
  Assessment of activities of daily living - no score just tick the box that applies; 'Not at all', 'With help', 'On your own with difficulty' and 'On your own'

CONTACTS AND LOCATIONS:
Overall Officials: Tom Wilkinson, Principal Investigator — Study Chief Investigator; Nick Francis, Principal Investigator — Study Deputy Chief Investigator
Locations (13):
- United Kingdom (13):
  - Belfast City Hospital, Belfast
  - Queen Elizabeth Hospital,, Birmingham
  - Bradford Royal Infirmary, Bradford
  - Park and St Francis Surgery, Chandler's Ford
  - Hull and East Yorkshire NHS Trust, Castle Hill Hospital,, Hull
  - Glenfield Hospital,, Leicester
  - Wythenshawe Hospital, Manchester
  - City Campus of Nottingham University, Nottingham
  - John Radcliffe Hospital, Oxford
  - The Adam Practice, Poole
  - The Virtual Team, Southampton
  - University Hospital Southampton Nhs Foundation Trust, Southampton
  - Oaks Healthcare, Waterlooville

IPD SHARING:
Plan to Share IPD: No
No plan to share data

REFERENCES:
- [Derived] Monk PD, Marsden RJ, Tear VJ, Brookes J, Batten TN, Mankowski M, Gabbay FJ, Davies DE, Holgate ST, Ho LP, Clark T, Djukanovic R, Wilkinson TMA; Inhaled Interferon Beta COVID-19 Study Group. Safety and efficacy of inhaled nebulised interferon beta-1a (SNG001) for treatment of SARS-CoV-2 infection: a randomised, double-blind, placebo-controlled, phase 2 trial. Lancet Respir Med. 2021 Feb;9(2):196-206. doi: 10.1016/S2213-2600(20)30511-7. Epub 2020 Nov 12. PMID 33189161
- [Derived] Lee JS, Shin EC. The type I interferon response in COVID-19: implications for treatment. Nat Rev Immunol. 2020 Oct;20(10):585-586. doi: 10.1038/s41577-020-00429-3. PMID 32788708